CLINICAL TRIAL: NCT04152577
Title: Lenalidomide, Rituximab and Combination Chemotherapy Versus Rituximab and Combination Chemotherapy in Treating Patients With Newly Diagnosed Highly Aggressive Non-Hodgkin B-cell Lymphoma
Brief Title: R2 and Combination Chemotherapy Versus R and Combination Chemotherapy in Newly Diagnosed Highly Aggressive B-NHL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Xin, Director of Hematology Department, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ShangdongPH
Record Dates: First submitted 2019-10-27; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Lymphoma, B-Cell
Keywords: Lenalidomide，rituximab，chemotherapy，highly aggressive B-NHL
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R2-combination chemotherapy (Experimental): R2-CHOP/CHOPE/DA-EPOCH/HD MTX
  R2-CHOP :
  lenalidomide 25mg/d po D1-10; Rituximab：375mg/m2，ivgtt，D0 Cyclophosphamide 750mg / m2 d1, doxorubicin 70mg / m2 or Doxorubicin liposome 30-40 mg / m2 d2, vincristine 1.4mg / m2 or vindesine 3mg / m2 d2, prednisone 100mg d1-5
  R2-DA-EPOCH:
  lenalidomide 25mg/d po D1-10; Rituximab：375mg/m2，ivgtt，D0 Epirubicin 15mg／m２ ,d1-4; Etoposide 50mg／m２ ,d1-4; Vincristine 0.4mg/ ｍ２ ，d1-4; Cyclophosphamide 750mg/ ｍ２ , d５; Prednisone 60mg/m２/d, d1-5;
  R2-HD MTX:
  lenalidomide 25mg/d po D1-10; Rituximab：375mg/m2，ivgtt，D0； MTX 3.5g／ｍ２,ｄ1
  Interventions: Drug: R2-combination chemotherapy
- R-combination chemotherapy (Active Comparator): R-CHOP/CHOPE/DA-EPOCH/HD MTX
  R-CHOP :
  Rituximab：375mg/m2，ivgtt，D0 Cyclophosphamide 750mg / m2 d1, doxorubicin 70mg / m2 or Doxorubicin liposome 30-40 mg / m2 d2, vincristine 1.4mg / m2 or vindesine 3mg / m2 d2, prednisone 100mg d1-5
  R-DA-EPOCH:
  Rituximab：375mg/m2，ivgtt，D0 Epirubicin 15mg／m２ ,d1-4; Etoposide 50mg／m２ ,d1-4; Vincristine 0.4mg/ ｍ２ ，d1-4; Cyclophosphamide 750mg/ ｍ２ , d５; Prednisone 60mg/m２/d, d1-5;
  R-HD MTX:
  Rituximab：375mg/m2，ivgtt，D0； MTX 3.5g／ｍ２,ｄ1
  Interventions: Drug: R-combination chemotherapy

INTERVENTIONS:
Drug: R2-combination chemotherapy — R2-CHOP/CHOPE/DA-EPOCH/HD MTX
  R2-CHOP :
  lenalidomide 25mg/d po D1-10; Rituximab：375mg/m2，ivgtt，D0 Cyclophosphamide 750mg / m2 d1, doxorubicin 70mg / m2 or Doxorubicin liposome 30-40 mg / m2 d2, vincristine 1.4mg / m2 or vindesine 3mg / m2 d2, prednisone 100mg d1-5
  R2-DA-EPOCH:
  lenalidomide 25mg/d po D1-10; Rituximab：375mg/m2，ivgtt，D0 Epirubicin 15mg／m２ ,d1-4; Etoposide 50mg／m２ ,d1-4; Vincristine 0.4mg/ ｍ２ ，d1-4; Cyclophosphamide 750mg/ ｍ２ , d５; Prednisone 60mg/m２/d, d1-5;
  R2-HD MTX:
  lenalidomide 25mg/d po D1-10; Rituximab：375mg/m2，ivgtt，D0； MTX 3.5g／ｍ２,ｄ1
  Arms: R2-combination chemotherapy
Drug: R-combination chemotherapy — R-CHOP/CHOPE/DA-EPOCH/HD MTX
  R-CHOP :
  Rituximab：375mg/m2，ivgtt，D0 Cyclophosphamide 750mg / m2 d1, doxorubicin 70mg / m2 or Doxorubicin liposome 30-40 mg / m2 d2, vincristine 1.4mg / m2 or vindesine 3mg / m2 d2, prednisone 100mg d1-5
  R-DA-EPOCH:
  Rituximab：375mg/m2，ivgtt，D0 Epirubicin 15mg／m２ ,d1-4; Etoposide 50mg／m２ ,d1-4; Vincristine 0.4mg/ ｍ２ ，d1-4; Cyclophosphamide 750mg/ ｍ２ , d５; Prednisone 60mg/m２/d, d1-5;
  R-HD MTX:
  Rituximab：375mg/m2，ivgtt，D0； MTX 3.5g／ｍ２,ｄ1
  Arms: R-combination chemotherapy

SUMMARY:
In this study，lenalidomide was added in the first-line treatment in the newly diagnosed highly invasively non-Hodgkin B-cell lymphoma. The R2-CHOP/R2-EPOCH etc was applied compared with the classical R-CHOP/R-EPOCH etc. The investigators tried to explore a more effective and safe treatment regimen for patients with high-risk B-cell lymphoma to improve the patient's poor prognosis.

DETAILED DESCRIPTION:
Lymphoma has become one of the top ten malignant tumors, of which non-Hodgkin's B-cell lymphoma accounts for the majority. As the classic first-line treatment, the emergence of the R-CHOP program has resulted in clinical cures for more than 1/2 of patients with B-cell lymphoma. But for patients with highly aggressively B cell lymphoma, most of them still suffer from disease recurrences due to R-CHOP treatment alone.

In recent years, with the emergence of various new drugs, many researchers have tried to add new drugs to the classic R-CHOP program as a first-line treatment for non-Hodgkin B-cell lymphoma. As a new type of immunomodulator, lenalidomide was first approved for the treatment of multiple myeloma. In recent years, its role in refractory and relapsed B-cell lymphoma has gradually been recognized.

In 2015, Nowakowski et al. published a clinical study of 64 patients with diffuse large B-cell lymphoma who used R2-CHOP in first-line therapy. It was found that R2-CHOP does not improve R-CHOP in patients with GCB. The effective rate of treatment and the 2-year survival rate of patients, but for patients with non-GCB type DLBCL with poor prognosis, the addition of lenalidomide can greatly improve the remission rate of the disease and improve the poor prognosis of patients.

So, the investigators initiate this study to evaluate the efficacy of R2-CHOP/R2-EPOCH etc in newly diagnosed highly invasively non-Hodgkin B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed highly aggressively B-Cell Non-Hodgkin's lymphoma (NHL) confirmed by histopathology
2. The patient has at least ≥1 measurable tumor lesion with a diameter >1.5 cm;
3. The patient has not undergone systemic chemotherapy or immunotherapy before;
4. ECOG score ≤ 2 points;
5. Liver and kidney function meets the following conditions: creatinine clearance rate ≥ 30ml / min, total bilirubin, AST and ALT ≤ 2.5 × ULN;
6. No history of malignant tumors within 5 years, except for cured carcinomas in situ such as basal cell carcinoma of the skin, cervical cancer, breast cancer, prostate cancer, etc.;
7. agree to take contraceptive measures during the trial period and within 3 months after the end of the trial;
8. Patients volunteered to participate in the study and signed informed consent.

Exclusion Criteria:

1. Serious cardiovascular and other important organs and blood, endocrine system lesions, and other history of malignant tumors;
2. Severe mental illness;
3. Pregnant or lactating women and men or women who intend to conceive in the near future;
4. The expected survival time is less than 6 months;
5. HBV, HCV or HIV infection or seropositive;
6. there are active infections;
7. Allergies or allergies to rituximab;
8. Compliance or poor follow-up;
9. Other circumstances that the investigator believes are not suitable for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-06-05 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate after 3 cycles | at the end of 3 cycles( each cycle is 21 days)
  Percentage of patients with complete remission （CR）or partial remission （PR）
Overall Response Rate after 6 cycles | at the end of 6 cycles( each cycle is 21 days)
  Percentage of patients with complete remission （CR）or partial remission （PR）

SECONDARY OUTCOMES:
Progression free survival（PFS） | 2 years
  Time from enrollment to tumor progression or death
overall survival（OS） | 2 years
  Time from enrollment to death

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wang, MD,PhD, Principal Investigator — Shandong Provincial Hospital
Locations (1):
- Department of Hematology, Provincial Hospital Affiliated to Shandong University, Jin'an, Shandong, China

IPD SHARING:
Plan to Share IPD: No